CLINICAL TRIAL: NCT04992039
Title: Evaluation of the WHO HEARTS Hypertension Control Package in the Primary Care Clinics of Bangladesh: A Quasi-experimental Trial
Brief Title: HEARTS Package Evaluation Trial in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Foundation of Bangladesh (Other)
Collaborators: Resolve to Save Lives (Other); National Heart Foundation Hospital and Research Institute, Bangladesh (Unknown); Non-communicable Disease Control Programme, Directorate General of Health Services, Bangladesh (Unknown); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: N.H.F.H.&R.I:4-14/7/AD/1074
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Hypertension; Hypertension Control Program; World Health Organization HEARTS Technical Package
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Equal number of participants will be recruited simultaneously in both group of control and intervention. After certain time period of intervention participants of both groups will be evaluated and the differences of outcome will be measured.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Participants of this arm will not receive the total WHO HEARTS package as an intervention. These participants will be screened in the designated area for universal BP screening via A&D arm-in device. Their diagnosis will be confirmed by measuring their BP by a Medical Officer via an Omron desktop oscillometer. The Medical Officers and UHC nurses of the control sites will be trained up on BP measurement using standard techniques, patient registration, data collection, etc.
- Intervention Arm (Experimental): Participants of this arm will receive all the components of WHO HEARTS technical package components as an intervention.
  Interventions: Other: WHO HEARTS technical package

INTERVENTIONS:
Other: WHO HEARTS technical package — Components of WHO HEARTS technical package are
  1. Universal BP screening via A&D arm-in BP device.
  2. Training of Medical Officers and Nurses on BP measurement using standard techniques.
  3. Training of the nurses on screening, registration data collection via the Simple mobile smart-phone digital clinical hypertension information application.
  4. Use of a drug and dose specific hypertension treatment protocol.
  5. Standardized inventory and procurement practice to ensure a reliable supply of protocol medications.
  6. Training and support for team-based model of hypertension care delivery.
  7. Access to the Simple data dashboard for program monitoring.
  8. Standardized procedure for patient follow-up.
  9. Community-based prescription refilling.
  Arms: Intervention Arm

SUMMARY:
Hypertension became the leading risk factor of death globally as well as in Bangladesh. Uncontrolled hypertension is the key challenge for the success of a hypertension control programs. According to the last national STEPS Survey in Bangladesh, hypertension control rate is only 11%. World Health Organization promoted the HEARTS technical package for the hypertension control programs to improve the control scenario. National Heart Foundation of Bangladesh is implementing a hypertension control program in selected Upazilas (sub-districts) of Bangladesh in collaboration with Non-Communicable Disease Control (NCDC) Program of Directorate General of Health Services (DGHS) and Resolve to Save Lives, USA. Proposed quasi experimental study will be conducted in collaboration with NCDC of DGHS, Resolve to Save Lives, USA and Johns Hopkins University, Baltimore with an objective of to evaluate the impact of HEARTS package on the rate of hypertension control in primary health care centers in Bangladesh. In this study equal number of hypertensive adult patients will be recruited in Upazila Health Complexes of control and intervention groups with a hypothesis of, implementation of HEARTS technical package in primary health care centers can reduce the blood pressure significantly. After obtaining informed written consent, respondents' basic demographic information, history of antihypertensive medication intake and related comorbidities will be taken. Blood pressure measurements data will be recorded also. All of these data will be collected via a secured mobile application, Simple App. Collected data will be preserved in a secured cloud based database. After six months of enrolment, and end-line data will be collected at the community setup, preferably at the home of respondents, following standard techniques of BP measurement by experienced Field Research Assistants. During whole of the study procedure, every ethical right of the participants will be preserved with an utmost priority. De-identified data will be shared with the partner organizations for further scientific analysis. This study will generate robust evidence for use of HEARTS technical packages in low-and middle-income countries, like Bangladesh, especially at low-level health facilities and provide guidance for designing and implementation of other hypertension control programs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Have a diagnosis of hypertension (inclusive of known prior diagnosis or a new diagnosis), with a baseline systolic BP ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg
* Eligible for the HEARTS technical package, i.e., are not pregnant, not being treated for an acute illness or medical emergency, and do not have a terminal illness.

Exclusion Criteria:

* Previously diagnosed hypertensive patients with a controlled BP at the time of enrollment (systolic BP <140 mmHg and diastolic BP < 90 mmHg). Either BP is controlled using diet and lifestyle measures or BP is controlled on antihypertensive medications,
* Cognitive impairment that would prevent comprehension of and responding to questions
* Patients who otherwise meet inclusion criteria but decline to participate in the hypertension program evaluation or are not able to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3935 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Difference in differences of systolic blood pressure (SBP) | Six months
  defined as between- group difference in BP change at six months (BP change at six months calculated for each group as end-line minus baseline mean systolic BP)

SECONDARY OUTCOMES:
Difference in differences of diastolic blood pressure (DBP) | Six months
  defined as between- group difference in BP change at six months (BP change at six months calculated for each group as end-line minus baseline mean diastolic BP)
Difference in differences of rate of hypertension control. | Six months
  defined (per UHC) as: NUMERATOR: Enrolled patients with controlled BP (SBP <140 and DBP <90 mmHg) measured in the community at six months/DENOMIN'ATOR: Total enrolled patients
Rate of loss to follow-up. | Six months
  defined (per UHC) as - NUMERATOR: Enrolled patients with no clinic visit in the 3 months previous to the six-month follow up/DENOMINATOR: Total enrolled patients
Difference in differences of rate of hypertension control (Measured in the clinic) | Six months
  defined (per UHC) as: NUMERATOR: Enrolled patients with controlled BP (SBP <140 and DBP <90 mmHg) at the most recent clinical visit within the 3 months previous to the six-month follow up/DENOMINATOR: Total enrolled patients
Rate of loss to follow up | Six months
  defined (per UHC) as: NUMERATOR: Enrolled patients with no clinic visit in the 3 months previous to the six-month follow up/DENOMINATOR: Total enrolled patients
Difference in time to BP control | Six months
  difference in time-to-control between arms based on follow-up in-clinic BP and assessed using the log-rank test

CONTACTS AND LOCATIONS:
Overall Officials: Sohel R Choudhury, PhD, Principal Investigator — National Heart Foundation Hospital and Research Institute
Locations (14):
- Bangladesh (14):
  - Madarganj Upazila Health Complex, Jāmālpur, Dhaka Division
  - Baniachang Upazila Health Complex, Habiganj
  - Madhabpur Upazila Health Complex, Habiganj
  - Bakhshiganj Upazila Health Complex, Jamālpur
  - Dewanganj Upazila Health Complex, Jamālpur
  - Islampur Upazila Health Complex, Jamālpur
  - Melandaha Upazila Health Complex, Jamālpur
  - Sarishabari Upazila Health Complex, Jamālpur
  - Karimganj Upazila Health Complex, Kishoreganj
  - Katiadi Upazila Health Complex, Kishoreganj
  - Tarail Upazila Health Complex, Kishoreganj
  - Biswamvarpur Upazila Health Complex, Sunāmganj
  - Doarabajar Upazila Health Complex, Sunāmganj
  - Gowainghat Upazila Health Complex, Sylhet

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared with the other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of data collection, deidentified IPD will be shared with the collaborators and those will be available for them till completion of the report writeup.
Access Criteria: IPD will be shared will the collaborator researchers who will participate in the data analysis and report writing.

REFERENCES:
- [Background] Mills KT, Bundy JD, Kelly TN, Reed JE, Kearney PM, Reynolds K, Chen J, He J. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation. 2016 Aug 9;134(6):441-50. doi: 10.1161/CIRCULATIONAHA.115.018912. PMID 27502908
- [Background] Kaur P, Kunwar A, Sharma M, Mitra J, Das C, Swasticharan L, Chakma T, Dipak Bangar S, Venkatasamy V, Dharamsoth R, Purohit S, Tayade S, Singh GB, Bitragunta S, Durgad K, Das B, Dar S, Bharadwaj R, Joshi C, Bharadwaj V, Khedkar S, Chenji S, Reddy SK, Sreedhar C, Parasuraman G, Kasiviswanathan S, Viswanathan V, Uike P, Gaigaware P, Yadav S, Dhaliwal RS, Ramakrishnan S, Tullu FT, Bhargava B. India Hypertension Control Initiative-Hypertension treatment and blood pressure control in a cohort in 24 sentinel site clinics. J Clin Hypertens (Greenwich). 2021 Apr;23(4):720-729. doi: 10.1111/jch.14141. Epub 2020 Dec 23. PMID 33369074
- [Background] Bloom DE, Cafiero E, Jané-Llopis E, Abrahams-Gessel S, Bloom LR, Fathima S, Feigl AB, Gaziano T, Hamandi A, Mowafi M, O'Farrell D. The global economic burden of noncommunicable diseases. Program on the Global Demography of Aging; 2012 Jan.
- [Background] World Health Organization. National STEPS survey for non-communicable diseases risk factors in Bangladesh 2018.
- [Background] World Health Organization. HEARTS Technical package for cardiovascular disease management in primary health care. Geneva: WHO; 2016.
- [Derived] Abrar A, Hu X, Akhtar J, Jubayer S, Noor Nabi Sayem M, Sultana S, Al Mamun MA, Bhuiyan MR, Malik F, Amin MR, Alim A, Gupta R, Zhao D, Farrell M, Banigbe B, Matsushita K, Burka D, Appel L, Moran AE, Choudhury SR. Evaluation of the World Health Organization-HEARTS hypertension control package in Bangladesh: a quasi-experimental trial. Heart. 2024 Aug 14;110(17):1090-1098. doi: 10.1136/heartjnl-2024-324253. PMID 39019496